CLINICAL TRIAL: NCT05200624
Title: Subthreshold Laser Treatment in Intermediate Age-related Macular Degeneration With Nascent Geographic Atrophy Study
Acronym: LIANA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with meeting recruitment targets
Sponsor: Center for Eye Research Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIANA
Record Dates: First submitted 2021-12-09; First posted 2022-01-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-06

CONDITIONS: Age-Related Macular Degeneration
Keywords: Laser; Subthreshold nanosecond laser; Nascent geographic atrophy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active laser (Active Comparator): Application of the active 2RT sub threshold laser
  Interventions: Device: 2RT subthreshold nanosecond laser
- Sham laser (Sham Comparator): Application of sham laser (i.e. flashing lights which replicate the look of active laser to the participant)
  Interventions: Device: 2RT subthreshold nanosecond laser

INTERVENTIONS:
Device: 2RT subthreshold nanosecond laser — The 2RT™ Q-switched YAG laser (532nm) delivering 3 nanosecond pulses; 400 um spot size, is a pulsed subthreshold nanosecond (SNL) laser, which uses low energy levels to produce limited effects that selectively target melanosomes within the pigmented retinal pigment epithelial (RPE) cells.
  Other Names: 2RT; SNL

SUMMARY:
This study is a prospective, single centre, randomized, sham-controlled, double-masked, clinical trial which aims to investigate the effect of subthreshold nanosecond laser on disease progression in eyes with intermediate age-related macular degeneration (AMD) and nascent geographic atrophy by functional and anatomical outcomes.

The study population will be individuals with high-risk intermediate age-related macular degeneration who meet all eligibility criteria. 60 subjects total (30 randomized to receive subthreshold nanosecond laser (SNL) treatment and 30 to receive sham treatment as per the 1:1 randomization).

The study has a 12-month study period with four scheduled visits: screening, randomisation (first treatment), 6-month follow up visit (with second treatment where eligible), 12-month follow-up.

The primary outcome is the proportion of laser-treated study eyes that develop late AMD compared to sham-treated study eyes over 12 months. The key secondary outcome is the change in retinal function of laser-treated study eyes compared to sham-treated study eyes over 12 months. Safety will be the proportion of laser-treated eyes that lose 10+ letters of vision (measured on a standard vision chart) compared to sham-treated eyes over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years or older at time of consent
2. Best corrected visual acuity (BCVA) of 59 letters (Snellen equivalent of 6/19) or better in both eyes
3. Bilateral large (>125µm) drusen as seen on colour fundus photographs (CFP) as assessed within a circle with radius of 3000µm centred on the fovea
4. Between 1 to 5 (inclusive) discrete area/s of nascent geographic atrophy (nGA) as seen on SD-OCT B-scan/s within a 20°x20° volume scan centred on the fovea in the study eye NOTE: TThe non-study eye does not need to have nGA but can have: any number of nGA, iRORA or cRORA lesions (on OCT) but not GA (on CFP or FAF)
5. Ability, willingness and sufficient cognitive awareness to consent to the trial, received randomized SNL treatment or sham procedure, and complete all visits as per the study schedule

Exclusion Criteria:

1. STUDY EYE: A cluster of definitely present reticular pseudodrusen (RPD) of >1 disc area (DA) (i.e., an area approximately 2.54mm2 in size) as seen on near infrared (NIR) imaging, or fundus autofluorescence (FAF) within a 20˚x20˚ field centred on the fovea
2. STUDY EYE: A subfoveal pigment epithelial detachment (PED)/drusenoid detachment >1000µm in diameter (measured on the central B-scan) with hyperreflective foci (HRF) and increased choroidal transmission or any PED >2000µm measured at the central foveal B-scan
3. Any evidence of definite geographic atrophy (GA) in either eye
4. Any evidence of active, regressed or treated macular neovascularization (MNV), in either eye, or active peripapillary CNV in the study eye (determined on multi-modal imaging and a fundus fluorescein angiogram is only required if in the investigator's medical judgement) NB: Subretinal fluid (SRF) <100µm or SRF associated with a subfoveal pseudovitelliform lesion permitted (i.e. slither/draping/ vitelliform with no evidence of new vessels on OCT-A) is not considered MNV and can be enrolled.
5. Any other investigational treatment for AMD, excluding dietary supplements, received in the past 12 months or thought, in the opinion of the investigator, likely to chronically change the course of the subject's retinal disease
6. Current participation in any other investigational ophthalmological clinical trial
7. Any ocular disease in the study eye, other than AMD, which in the opinion of the investigator may significantly compromise assessment of the retina, or which would compromise the ability to assess any effect following SNL treatment including, but not limited to:

   1. Diabetic retinopathy (unless limited to fewer than 10 microaneurysms and/or small retinal hemorrhages, without retinal thickening on OCT)
   2. Macular pathology or pigmentary abnormalities atypical of AMD, including but not limited to: pattern dystrophy, myopic maculopathy, angioid streaks, resumed ocular histoplasmosis syndrome, central serous choroidopathy, visually-significant epiretinal membranes, macular hole or pseudohole
   3. Optic nerve pathology, including optic atrophy, history of optic neuropathy
   4. Myopic crescent wider than 50% of the longest diameter of the optic disc, or closer than 1500 µm to the fovea
   5. Retinal vascular diseases including branch or central vein or artery occlusion
   6. Choroidal nevus within 2 disc diameters (DD) of the fovea associated with depigmentation or overlying drusen, if these drusen are used to determine eligibility
   7. Active uveitis or ocular inflammation
8. History or presence of uncontrolled glaucoma
9. Intraocular pressure which would preclude safe dilation of the pupil to allow adequate assessment and application of SNL treatment
10. History of prior laser surgery to the retina including subthreshold laser (focal retinopexy for a peripheral break and/or focal retinal tears performed more than 90 days prior to the entry into the study is permitted)
11. Significant cataract or other ocular media which, in the opinion of the investigator, significantly limits the visual acuity or view of the retina
12. Previous retinal or ocular surgery, the effects of which may now or in the future complicate assessment of the progression of AMD. (Cataract surgery is allowed as long as it was performed over 90 days prior to entry into the study)
13. Known hypersensitivity to fluorescein
14. Sensitivity to application of a contact lens
15. Corneal pathology precluding visualization of fundus or increasing the risk of using a contact lens, such as corneal dystrophy, recurrent corneal erosion syndrome or sensitivity to the application of a contact lens.
16. Use of any systemic or ocular medication known to be toxic to the retina, excluding tamoxifen unless there is evidence of toxicity.
17. Pregnant or lactating women
18. Subject who is considered ineligible for this study in the investigator's medical judgement

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Rate of progression to advanced AMD in study eyes | 12 months
  The time to develop advanced AMD - as defined as choroidal neovascularization (CNV), geographic atrophy (GA), or OCT-defined cRORA - in the SNL-treated compared to sham-treated study eyes over 12 months

SECONDARY OUTCOMES:
Rate of retinal sensitivity change in study eyes | 12 months
  The rate of change in mean retinal sensitivity over time (in decibels per year) of the SNL-treated compared to sham-treated study eyes over 12 months.

OTHER OUTCOMES:
Safety Endpoint: Proportion of study eyes with a ≥10-letter loss in best-corrected visual acuity (BCVA) | 12 months
  The proportion of eyes that lose ≥10 letters of BCVA in the SNL-treated compared to sham-treated study and fellow eyes over 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn H Guymer, MBBS FRANZCO, Principal Investigator — Center for Eye Research Australia
Locations (4):
- Australia (4):
  - Marsden Eye Specialists, Parramatta, New South Wales
  - Adelaide Eye & Retina Centre, Adelaide, South Australia
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Retinology Institute, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No